CLINICAL TRIAL: NCT02091505
Title: Predictive Factors of Treatment Outcome After Intravitreal Injection of Lucentis (Ranibizumab) in Eyes With Macular Edema Associated With Central Retinal Vein Occlusion (CRVO)
Brief Title: Predictive Factors of Ranibizumab Treatment in Macular Edema With CRVO
Acronym: CRVO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mie University (Other)
Responsible Party: Principal Investigator, Mineo Kondo, MD. PhD., Mie University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MKONDO-CRVO
Record Dates: First submitted 2014-03-16; First posted 2014-03-19 (Estimated); Last update posted 2014-03-19 (Estimated); Status verified 2014-03

CONDITIONS: Central Retinal Vein Occlusion
MeSH Terms: conditions — Retinal Vein Occlusion | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intravitreal injection of Ranibizumab (Experimental)
  Interventions: Drug: Ranibizumab

INTERVENTIONS:
Drug: Ranibizumab

SUMMARY:
Recent studies have shown that intravitreal injection of anti-VEGF agent, Lucentis (Ranibizumab) is effective for macular edema associated with central retinal vein occlusion (CRVO). However, there is little information on whether there are any predictive factors of treatment outcome after this treatment. We plan to perform comprehensive functional and imaging tests to determine significant predictive factors.

DETAILED DESCRIPTION:
The purpose of the present study is to investigate predictive factors of treatment outcome after intravitreal injection of Lucentis (Ranibizumab) in eyes with macular edema associated with central retinal vein occlusion (CRVO) using various comprehensive clinical tests including visual filed, spectral-domain optical coherence tomography (SD-OCT), ultra wide-field fluorescein angiography, new flicker electroretinogram (ERG) using skin electrodes. Corrected visual acuity, visual filed, spectral-domain optical coherence tomography (SD-OCT), ultra wide-field fluorescein angiography, and new flicker electroretinogram (ERG) using skin electrodes are performed before and 3, 6, 9, 12 months after the treatment. Predictive factors of treatment outcome are statistically analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Macular edema associated with central retinal vein occlusion
* Best corrected visual acuity < 20/30
* Central macular thickness > 300
* Period from symptom onset to treatment < 12 months

Exclusion Criteria:

* Any past history of treatment for macular edema (e.g. anti-VEGF injection, steroid, vitrectomy)

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-12; Primary Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Best-corrected visual acuity | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Mineo Kondo, MD, PhD, Study Director — Mie University Hospital
Locations (1):
- Mie University Hospital, Tsu, Aichi-ken, Japan

REFERENCES:
- [Background] Brown DM, Campochiaro PA, Singh RP, Li Z, Gray S, Saroj N, Rundle AC, Rubio RG, Murahashi WY; CRUISE Investigators. Ranibizumab for macular edema following central retinal vein occlusion: six-month primary end point results of a phase III study. Ophthalmology. 2010 Jun;117(6):1124-1133.e1. doi: 10.1016/j.ophtha.2010.02.022. Epub 2010 Apr 9. PMID 20381871
- [Background] Bhisitkul RB, Campochiaro PA, Shapiro H, Rubio RG. Predictive value in retinal vein occlusions of early versus late or incomplete ranibizumab response defined by optical coherence tomography. Ophthalmology. 2013 May;120(5):1057-63. doi: 10.1016/j.ophtha.2012.11.011. Epub 2013 Feb 14. PMID 23415775
- See also: Department of Ophthalmology, Mie University Graduate School of Medicine — http://www.medic.mie-u.ac.jp/ophthalmology/